CLINICAL TRIAL: NCT04428983
Title: The Effect of Hericium Erinaceus Mycelium in Non-motor Symptoms of Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Yuan-Ting Sun, Doctor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HELPD V4 20191120
Record Dates: First submitted 2019-11-20; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease, non-motor symptoms
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hericium erinaceus mycelium (Experimental): Hericium erinaceus capsules 1 table tid orally per day for 24 months
  Interventions: Dietary Supplement: Hericium erinaceus mycelium
- placebo (Placebo Comparator): placebo capsules 1 table tid orally per day for 24 months
  Interventions: Dietary Supplement: Hericium erinaceus mycelium

INTERVENTIONS:
Dietary Supplement: Hericium erinaceus mycelium — Hericium erinaceus capsules 3 tables per day for 24 months

SUMMARY:
Parkinson disease (PD) is considered a multisystemic neurodegenerative disorder, together with the classic motor disability, and a number of non-motor symptoms (NMS).NMS have a significant negative relation with patients' quality of life. In general, both medicinal and nonmedicinal therapies are often advised for PD patients with NMS, but robust evidences for underpinning the clinical effects are limited. Recently, the search for small preventative neurotrophic compounds that are responsible for the maintenance, survival of neurons has attracted much attention. Erinacine A, which is extracted from Hericium erinaceus is the one showed prominent beneficial effects in the central nervous system. It can increase NGF and catecholamine content in the locus coeruleus and hippocampus of rats. This markedly increases neuronal survival in different brain areas and substantially improve behavioral outcomes in various animal models. In a MPTP-induced Parkinsonism model, treatment with Hericium erinaceus mycelium reduced the loss of dopaminergic cell, eliminated neuronal apoptosis and reversed MPTP-associated motor deficits. Thus, this project intends to hold a randomized, controlled trial to assess the effect of Hericium erinaceus mycelium, which is enriched of Erinacine A, in NMS of PD. This project will enroll 80 patients with PD. Subjects will be randomly allocated into study or placebo group. Subjects will take Hericium erinaceus mycelium for 2 years (one capsule per meal per day) and their treatments for PD will not be altered.

DETAILED DESCRIPTION:
Inclusion criteria:

1. PD patients aged 50-79 years diagnosed by neurologist (should exclude vascular parkinsonism, secondary parkinsonism( including toxin, drug, heavy metal, CO intoxication), normal pressure hydrocephalus, multiple system atrophy, progressive supranuclear palsy, cortical basal degeneration, dementia with Lewy Body, hereditary parkinson's disease with genetic mutation, Huntington's disease, Wilson disease, spinal cerebellar ataxia with extrapyramidal syndrome, essential tremor, dystonia)
2. PD at Hoehn and Yahr stage 2-2.5
3. without cognitive decline

Exclusion criteria:

1. with diabetes mellitus (DM)
2. with nephropathy (GFR < 30ml/min)
3. with significant neurological deficits caused by vascular insults

Measurement parameters:

1. At recruitment: blood sugar, AST, ALT, BUN, Crea, Ca, Na, K and peripheral blood cell (for the expression levels of KATP)
2. every 6 months: motor symptoms: UPDRS, evaluate with UDYSRS if presence with dyskinesia Non motor symptoms: self-report: PDQ39, QUIP, PDSS Rated by neurologist: NMSS, HAM-D, BPRS
3. every 1 year: CASI, tilting table, AST, ALT, BUN, crea, Na, K, Ca

Protocol:

0 month (initial baseline):

1. blood sugar, AST, ALT, BUN, Crea, Ca, Na, K and peripheral blood cell
2. Tilting table test (autonomic function)
3. CASI cognitive test
4. UPDRS, evaluate with UDYSRS if presence with dyskinesia Non motor symptoms: self-report: PDQ39, QUIP, PDSS Rated by neurologist: NMSS, HAM-D, BPRS
5. stool microbiota

6 months: UPDRS, evaluate with UDYSRS if presence with dyskinesia Non motor symptoms: self-report: PDQ39, QUIP, PDSS Rated by neurologist: NMSS, HAM-D, BPRS

12 months:

1. UPDRS, evaluate with UDYSRS if presence with dyskinesia Non motor symptoms: self-report: PDQ39, QUIP, PDSS Rated by neurologist: NMSS, HAM-D, BPRS
2. CASI cognitive test, tilting table, AST, ALT, BUN, crea, Na, K, Ca

18 months: UPDRS, evaluate with UDYSRS if presence with dyskinesia Non motor symptoms: self-report: PDQ39, QUIP, PDSS Rated by neurologist: NMSS, HAM-D, BPRS

24 months:

1. UPDRS, evaluate with UDYSRS if presence with dyskinesia Non motor symptoms: self-report: PDQ39, QUIP, PDSS Rated by neurologist: NMSS, HAM-D, BPRS
2. CASI cognitive test, tilting table, AST, ALT, BUN, crea, Na, K, Ca
3. stool microbiota

ELIGIBILITY:
Inclusion Criteria:

* idiopathic PD patients, aged 50-79 years
* modified Hoehn & Yahr stage 2-2.5
* Without subjective and objective cognitive decline (objective cognitive decline will be determined by CASI)

Exclusion Criteria:

* With diabetes
* With end stage renal disease under hemodialysis
* With significant vascular insults that resulted in significant neurological deficits

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2022-03-20 (Estimated); Study Completion 2023-03-20 (Estimated)

PRIMARY OUTCOMES:
baseline | 0 month
  Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
1st | 6 momths
  Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
2nd | 12 months
  Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
3rd | 18 months
  UPDRS
final | 24 months
  Unified Parkinson's Disease Rating Scale (MDS-UPDRS)

CONTACTS AND LOCATIONS:
Overall Officials: Li-Ya Lee, Study Director — Bioengineering Center, Grape King Bio
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided